CLINICAL TRIAL: NCT03931694
Title: Evaluation of the Feasibility of an E-health Tool in the Follow-up and Characterization of Chronic Pain Patients.
Brief Title: E-health Tool for Management of Chronic Pain Patients.
Acronym: e-DOL
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Institut ANALGESIA (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHU-425; 2018-A01790-5546 (Other: 2018-A01790-5546)
Record Dates: First submitted 2019-02-07; First posted 2019-04-30 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Chronic Pain
Keywords: Chronic pain; e-Health
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients with chronic pain follow in pain clinic
  Interventions: Device: e-DOL

INTERVENTIONS:
Device: e-DOL — e-health program (smartphone and web platform)

SUMMARY:
Chronic pain affects approximately 20% of adults, 50% of the elderly population and over 1.5 billion people worldwide. Societal and economic issues are also crucial, as 60% of people with pain are less able or unable to work and 20% say they have lost their jobs because of pain. The overall cost of chronic pain is estimated at around 300 billion euros in the EU. Unfortunately, current treatments for chronic pain have limited effectiveness. Pain clinics, which support the most complex and refractory cases of chronic pain, as well as general practitioners and patients expect improvements, both in terms of therapeutic efficacy and organization of care.

In order to allow the characterization and a personalized follow-up of chronic pain patients, Investigator has created e-DOL, a smartphone application for patients and a web platform for physicians. The purpose of this study is to evaluate the feasibility and clinical interest of an e-Health smartphone application for the characterization and follow-up of chronic pain patients..

DETAILED DESCRIPTION:
This first clinical study will assess the acceptability of the tool both by caregivers at the 13 pain clinics and by a panel of 300 patients followed for 6 months. Based on the results of the study (end 2019), investigator will improve the tool in a version 2.0, which will then be evaluated in a large impact study, measuring the intrinsic therapeutic effect of eDOL.

ELIGIBILITY:
Inclusion Criteria:

* All patients with chronic pain
* patients with and regular users of a smartphone
* Non-opposition to participation in the study

Exclusion Criteria:

* Patient unable to understand or answer questionnaires

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic pain
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
Feasibility of the e-health tool | Once, up to 12 months
  Feasibility evaluated by analysis of user acceptability (custom questionnaire: ease of use, utility...)
Feasibility of the e-health tool | Once, up to 12 months
  Feasibility evaluated by analysis of Number of data completed / missing (% of responses)
Feasibility of the e-health tool | Once, up to 12 months
  Feasibility evaluated by analysis of Participation of investigator centres (inclusion rate)

SECONDARY OUTCOMES:
Typology of patient responses | Weekly, up to 6 months
  Temporal evolution of the pain intensity using 0-10 VAS
Typology of patient responses | Up to 6 months
  Temporal evolution of the anxiety using 0-10 VAS
Typology of patient responses | Up to 6 months
  Temporal evolution of the sleep quality using 0-10 VAS
Typology of patient responses | Up to 6 months
  Temporal evolution of the mood using 0-10 VAS
Typology of patient responses | Up to 6 months
  Temporal evolution of the body comfort using 0-10 VAS
Typology of patient responses | Up to 6 months
  temporal evolution of the chronic pain symptoms and related-comorbidities by Brief Pain Inventory questionnaire
Typology of patient responses | Up to 6 months
  temporal evolution of the chronic pain symptoms and related-comorbidities by Pain Beliefs and Perceptions Inventory questionnaire
Typology of patient responses | Up to 6 months
  temporal evolution of the chronic pain symptoms and related-comorbidities by Medical Outcomes Study-Sleep Scale questionnaire
Typology of patient responses | Up to 6 months
  temporal evolution of the chronic pain symptoms and related-comorbidities by Tampa Scale of Kinesiophobia questionnaire
Typology of patient responses | Up to 6 months
  temporal evolution of the chronic pain symptoms and related-comorbidities by Pain Catastrophizing Scale questionnaire
Typology of patient responses | Up to 6 months
  temporal evolution of the chronic pain symptoms and related-comorbidities by EQ-5D questionnaire
Typology of patient responses | Up to 6 months
  temporal evolution of the chronic pain symptoms and related-comorbidities by ,Hospital Anxiety Depression Scale questionnaire
impact of the eHealth tool | Once, Up to 12 months.
  evaluation of the impact of the eHealth tool on current practices (clinician's opinion)
impact of the eHealth tool | Once, up 12 months.
  evaluation of the impact of the eHealth tool on quality of life (patient's opinion)

CONTACTS AND LOCATIONS:
Overall Officials: Noémie DELAGE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (13):
- France (13):
  - Chu Amiens, Amiens
  - Ch Bayeux, Bayeux
  - Chu Clermont-Ferrand, Clermont-Ferrand
  - Chu Grenoble, Grenoble
  - Chu Limoges, Limoges
  - Hospices Civils de Lyon, Lyon
  - Chu Nimes, Nîmes
  - AP-HP Ambroise Paré, Paris
  - Ap-Hp Cochin, Paris
  - Ap-Hp Lariboisiere, Paris
  - Chu Rouen, Rouen
  - Chu Toulouse, Toulouse
  - Ch Voiron, Voiron

REFERENCES:
- [Derived] Kerckhove N, Delage N, Cambier S, Cantagrel N, Serra E, Marcaillou F, Maindet C, Picard P, Martine G, Deleens R, Trouvin AP, Fourel L, Espagne-Dubreuilh G, Douay L, Foulon S, Dufraisse B, Gov C, Viel E, Jedryka F, Pouplin S, Lestrade C, Combe E, Perrot S, Perocheau D, De Brisson V, Vergne-Salle P, Mertens P, Pereira B, Djiberou Mahamadou AJ, Antoine V, Corteval A, Eschalier A, Duale C, Attal N, Authier N. eDOL mHealth App and Web Platform for Self-monitoring and Medical Follow-up of Patients With Chronic Pain: Observational Feasibility Study. JMIR Form Res. 2022 Mar 2;6(3):e30052. doi: 10.2196/30052. PMID 35234654